CLINICAL TRIAL: NCT04082156
Title: The Effect of Transcutaneous Electrical Nerve Stimulation on People With Muscle Fatigue Due to Training, Sports
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Omron Healthcare Co., Ltd. (Industry)
Collaborators: Western Michigan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HI794-0014
Record Dates: First submitted 2019-08-28; First posted 2019-09-09 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Muscle Fatigue
Keywords: TENS, DOMS, soreness, fatigue
MeSH Terms: conditions — Fatigue | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active TENS (Active Comparator)
  Interventions: Device: electrical stimulation
- Sham TENS (Sham Comparator)
  Interventions: Device: Sham

INTERVENTIONS:
Device: electrical stimulation — electrical stimulation
  Arms: Active TENS
Device: Sham — no stimulation
  Arms: Sham TENS

SUMMARY:
The objective is to assess if TENS will improve the muscle recovery rate from post-exercise fatigue.

ELIGIBILITY:
Inclusion Criteria:

* No phobia of electrical stimulation
* No pain or anti-inflammatory medication will be taken during study
* English speaking

Exclusion Criteria:

* Pregnancy
* Diabetes Mellitus
* Neuropathy
* Smoker
* Uncontrolled Hypertension
* Past surgery in the region to be treated by TENS or had received an intra-articular corticosteroid or hyaluronic acid injection within 6 months prior to enrollment
* Rhumatoid Arthritis (RA) in the area to be treated by TENS
* Allergic to tape/electrodes
* Dementia
* History of knee joint replacement or tibial osteotomy
* Undergoing physical therapy
* Any major joint pain (e.g., back, hip, or ankle) that could limit functional ability
* Contraindications to TENS such as having a pacemakers, dermatological conditions, and abnormal sensation of the lower extremity.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
VAS(Visual Analog Scale score) for soreness or pain | 2weeks
  Participants will record their level of knee pain by drawing a vertical mark between the ends of a 10-cm horizontal line. The 0-cm end and the 10-cm end represented no pain and the most extreme pain, respectively. The distance from the 0-cm end to the drawn mark was recorded to the first decimal place.
FI (Fatugue Index) | 2weeks
  A system called "Just Jump" by Probotics* will be used to induce DOMS. The goal of the jump is to create fatigue of the lower extremities which is a byproduct of decreased power. It will also create exercise induces DOMS. Using this system the next day will test the fatigue and power of the lower extremities to see if it has changed.

SECONDARY OUTCOMES:
sleep quality measurement | 2weeks
  Each subject will be provided with Sleep measurment device. The device captures sleep data via a sensor to monitor breathing, body movemement along with ambient light and temperature in the bedroom. The device is composed of six sleep parameters that combine to reflect the overall quality of sleep. It has objective sleep data, SleepScore (Objective Sleep Quality), MindScore (Objective REM Sleep Quality), BodyScore (Objective Deep Sleep Quality), Total Record Time, Time in Bed, Total Sleep Time, REM Sleep Time, Light Sleep Time, Deep Sleep time, Onset Time, WASO, Total Wake Time, Interruptions.
POMS (Profile of Mood States) | 2weeks
  It will be used for mental alertness. It is short form containing 24 items and four scales. Used in sports science (along with other areas) to evaluate and access mood after exercise or a sporting event concerned the certain scales containing "vigour" and "fatigue".

CONTACTS AND LOCATIONS:
Locations (1):
- Omron healthcare Co.,Ltd., Mukō, Japan